CLINICAL TRIAL: NCT04289662
Title: A Multicenter, Open-label Study to Evaluate 52 Weeks Long Term Efficacy and Safety of K-924 in Patients With Hypercholesterolemia Who Were Treated With Pitavastatin 2 mg or 4 mg.
Brief Title: K-924 Phase III Long Term Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kowa Company, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K-924-03
Record Dates: First submitted 2020-02-26; First posted 2020-02-28 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- K-924 LD (Experimental): K-924 LD once daily
  Interventions: Drug: K-924 LD
- K-924 HD (Experimental): K-924 HD once daily
  Interventions: Drug: K-924 HD

INTERVENTIONS:
Drug: K-924 LD — Pitavastatin 2 mg / Ezetimibe 10 mg tables
  Arms: K-924 LD
Drug: K-924 HD — Pitavastatin 4 mg / Ezetimibe 10 mg tables
  Arms: K-924 HD

SUMMARY:
A Multicenter, Open-label Study to Evaluate 52 weeks long term Efficacy and Safety of K-924 in Patients with hypercholesterolemia who were treated with pitavastatin 2 mg or 4 mg.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with hypercholesterolemia had to be age 20 years or older at written informed consent (ICF)
2. Patients who have been on a diet and / or exercise regimen more than 4 weeks before the screening
3. Patients who have been receiving pitavastatin calcium 2 mg / day or pitavastatin calcium 4 mg / day at least 4 weeks prior to the screening
4. Those whose LDL-C (Friedewald formula) at the screening any of the following in the category classification based on Japan Atherosclerosis Society guidelines for prevention Atherosclerotic Cardiovascular Disease 2017

   * Low risk of primary prevention : LDL-C => 160 mg/dL
   * Medium risk of primary prevention : LDL-C => 140 mg/dL
   * High risk of primary prevention : LDL-C => 120 mg/dL
   * Secondary prevention patients with a history of coronary artery disease : LDL-C => 100 mg/dL
   * Secondary prevention patients with familial hypercholesterolemia or acute coronary syndrome, or diabetes with other high-risk conditions : LDL-C => 70 mg/dL

Exclusion Criteria:

1. Patients with a history of myopathy or rhabdomyolysis due to pitavastatin or ezetimibe
2. Patients with a history of hypersensitivity due to pitavastatin or ezetimibe
3. Patients with severe liver damage (Child Pugh Class B or higher) or biliary obstruction
4. Pregnant women, lactating women, women planning to become pregnant or lactating during the study period, or pregnant women who do not use specific contraceptive methods
5. Patients whose CK is 3 times or more of the upper limit of the reference value at screening
6. Patients whose AST and ALT is 2 times or more of the upper limit of the reference value at screening
7. Patients wiht type 1 diabetes or uncontrolled type 2 diabetes as defined HbA1c 8 % or more at screening
8. Patients with uncontrolled hypertension as defined systolic blood pressure of 160 mmHg or more or diastolic blood pressure of 100 mmHg or more at screening
9. Patients with eGFR of less than 30 mL / min / 1.73 m² at screening or dialysis
10. Patients with heart failure class III or higher according to NYHA cardiac function classification
11. Patients with uncontrolled arrhythmia
12. Patients with uncontrolled metabolic endocrine disease
13. Patients with malignant tumors or who are judged to have a high possibility of relapse
14. Patients who developed acute coronary syndrome or stroke within 12 months before obtaining consent
15. Patients who have collected 200 mL or more within 4 weeks before screening, 400 mL or more of blood within 12 weeks for males or 16 weeks for females, or within 2 weeks for (Plasma component / platelet component)
16. Persons with a history of severe drug allergy (anaphylactic shock, etc.)
17. Patients who need contraindicated drugs during the study period after obtaining consent
18. Patients with TG of 400 mg / dL or more at screening
19. Patients who have LDL apheresis
20. Patients with malabsorption or history, or who have undergone gastrointestinal surgery (excluding appendectomy, hernia treatment, etc.) that may affect absorption.
21. Patients with Alcohol or drug addiction
22. Patients who participate in other clinical trials within 16 weeks prior to study drug administration and who are administered non-placebo investigational drugs, or who participate in other clinical trials concurrently with this study
23. Patients who have received K-924
24. Patients who judged to be inappropriate by the Investigator or Investigator

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2020-03-23 (Actual); Primary Completion 2021-08-07 (Actual); Study Completion 2021-08-07 (Actual)

PRIMARY OUTCOMES:
Efficacy: % change from baseline in LDL-C (Friedewald formula) (mg/dL) | Week 52

SECONDARY OUTCOMES:
Efficacy: % change or change from baseline in LDL-C (mg/dL) | From baseline upto week 52
Efficacy: % change or change from baseline in non-HDL-C (mg/dL) | From baseline upto week 52
Efficacy: % change or change from baseline in HDL-C (mg/dL) | From baseline upto week 52
Efficacy: % change or change from baseline in Total Cholesterol (mg/dL) | From baseline upto week 52
Efficacy: % change or change from baseline in TG (mg/dL) | From baseline upto week 52

CONTACTS AND LOCATIONS:
Locations (13):
- Japan (13):
  - Chubu Rosai Hospital, Aichi
  - Daido Clinic, Aichi
  - Nakamura Cardiovascular Clinic, Fukuoka
  - Nippon Kokan Fukuyama Hospital, Hiroshima
  - Hasegawa Medicine Clinic, Hokkaido
  - Miyanomori Memorial Hospital, Hokkaido
  - Yuri Ono Clinic, Hokkaido
  - Ota General Hospital, Kanagawa
  - Suwa Red Cross Hospital, Nagano
  - Shiraiwa medical clinic, Osaka
  - Minamino Cardiovascular Hospital, Tokyo
  - Tokyo Shinagawa Hospital, Tokyo
  - Tokyo-Eki Center-building Clinic, Tokyo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ako J, Yokote K, Tsujita K, Tanigawa R, Kamei R, Suganami H. Long-term Efficacy and Safety of K-924 Pitavastatin/Ezetimibe Fixed-dose Combination in Patients with Hypercholesterolemia: A Phase III, Multi-center, Open-label Trial. J Atheroscler Thromb. 2024 Mar 1;31(3):288-305. doi: 10.5551/jat.64272. Epub 2023 Sep 16. PMID 37722882